CLINICAL TRIAL: NCT02594098
Title: A Pilot Study to Evaluate the Efficacy and Safety of Secukinumab in the Treatment of Moderate to Severe Atopic Dermatitis
Brief Title: Secukinumab for Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Emma.Guttman, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 15-1486; CAIN457AUS02T (Other: Novartis Pharmaceuticals Corporation)
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; extrinsic atopic dermatitis; intrinsic atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

ARMS (2):
- Secukinumab (Experimental): Secukinumab (300 mg) via subcutaneous injection using 2 prefilled syringes
  Interventions: Drug: Secukinumab
- Placebo (Placebo Comparator): Placebo via subcutaneous injection using 2 prefilled syringes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab — At Weeks 0, 1, 2, 3, 4 and every 2 weeks thereafter through and including Week 12 in phase 1 of the study.
  Arms: Secukinumab
Drug: Placebo — At Weeks 0, 1, 2, 3, 4 and every 2 weeks thereafter through and including Week 12 in phase 1 of the study.
  Arms: Placebo

SUMMARY:
Atopic Dermatitis, also known as atopic eczema, or eczema, is a common skin disease that can affect males and females of all ages, but often starts in childhood. Recent studies show at least 4-7% of adults and 15-25% of children to be affected, with one third of patients having severe disease. It results in very itchy, red, swollen, and cracked skin. Scratching worsens the symptoms and causes the skin to become thickened over time. Patients with atopic dermatitis have an increased risk of skin infections, and many also develop hay fever or asthma. Atopic dermatitis can cause significant distress to both patients and their families.

In this study, the aim is to assess the effects of a new treatment called secukinumab in patients with atopic dermatitis. A total of 30 patients will be included in the study, which will run for a total of 52 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, pilot study of a total of 44 subjects with AD (22 with intrinsic and 22 with extrinsic AD) consisting of 2 phases. Subjects will be randomized (2:1) to either receive secukinumab 300 mg or placebo via subcutaneous injection using 2 prefilled syringes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject at least 18 years of age
* If female, the subject is not pregnant or nursing
* Subject is able to provide written informed consent and comply with the requirements of this study protocol.
* Chronic (>6 months) atopic dermatitis (intrinsic disease with IgE levels that are below 200, and extrinsic disease with IgE levels above 200).
* Moderate to severe AD (SCORAD index ≥25, and IGA index≥3).
* Subjects who are women of childbearing potential must have a negative urine pregnancy test at screening and must be practicing an adequate, medically acceptable method of birth control for at least 30 days before Day 0 and at least 6 months after the last study drug administration. Acceptable methods of birth control include intrauterine device (IUD); oral, transdermal, implanted or injected hormonal contraceptives (must have been initiated at least 1 month before entering the study); tubal ligation; abstinence and barrier methods with spermicide. Otherwise, if not of childbearing potential, subjects must: have a sterile or vasectomized partner; have had a hysterectomy, a bilateral oophorectomy or be clinically diagnosed infertile; or be in a menopausal state for at least a year.
* Tuberculin purified protein derivative (PPD) or QuantiFERON TB-Gold test (QFT) negative at the time of screening, or if patient has a history of positive PPD or QuantiFERON, he/she has completed the appropriate prophylaxis.
* Subject is judged to be in good general health as determined by the principal investigator based upon the results of medical history, laboratory profile, and physical examination.
* Patients with stable chronic asthma, treated with inhaled corticosteroids, will be allowed to participate.

Exclusion Criteria:

* Male or female subject at least 18 years of age
* If female, the subject is not pregnant or nursing
* Subject is able to provide written informed consent and comply with the requirements of this study protocol.
* Chronic (>6 months) atopic dermatitis (intrinsic disease with IgE levels that are below 200, and extrinsic disease with IgE levels above 200).
* Moderate to severe AD (SCORAD index ≥25, and IGA index≥3).
* Subjects who are women of childbearing potential must have a negative urine pregnancy test at screening and must be practicing an adequate, medically acceptable method of birth control for at least 30 days before Day 0 and at least 6 months after the last study drug administration. Acceptable methods of birth control include intrauterine device (IUD); oral, transdermal, implanted or injected hormonal contraceptives (must have been initiated at least 1 month before entering the study); tubal ligation; abstinence and barrier methods with spermicide. Otherwise, if not of childbearing potential, subjects must: have a sterile or vasectomized partner; have had a hysterectomy, a bilateral oophorectomy or be clinically diagnosed infertile; or be in a menopausal state for at least a year.
* Tuberculin purified protein derivative (PPD) or QuantiFERON TB-Gold test (QFT) negative at the time of screening, or if patient has a history of positive PPD or QuantiFERON, he/she has completed the appropriate prophylaxis.
* Subject is judged to be in good general health as determined by the principal investigator based upon the results of medical history, laboratory profile, and physical examination.
* Patients with stable chronic asthma, treated with inhaled corticosteroids, will be allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-11; Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Secukinumab Extrinsic: Secukinumab (300 mg) via subcutaneous injection using 2 prefilled syringes at Weeks 0, 1, 2, 3, 4.
  Thereafter through Week 16, the first 36 patients assessed at baseline received secukinumab 300 mg Q4W, while the remaining 5 patients received a higher dosing schedule of secukinumab 300 mg Q2W.
  Starting at Week 16, all subjects received secukinumab 300 mg. Patients initially randomized to secukinumab 300 mg Q4W or the higher dosing secukinumab 300 mg Q2W continued to receive their respective dosages through Week 48.
- Placebo Then Secukinumab Extrinsic: Placebo via subcutaneous injection using 2 prefilled syringes at Weeks 0, 1, 2, 3, 4.
  Thereafter through Week 16, the first 36 patients assessed at baseline received placebo Q4W, while the remaining 5 patients received a higher dosing schedule of placebo Q2W.
  Starting at Week 16, all subjects received secukinumab 300 mg. Patients initially randomized to placebo Q4W or the higher dosing placebo Q2W received secukinumab 300 mg Q4W from Week 16 to Week 20, followed by every 4 weeks until Week 48 or every 2 weeks through Week 48 for the higher dosing schedule.
Period: Overall Study
Arm/Group | Secukinumab Extrinsic | Placebo Then Secukinumab Extrinsic
Started | 27 | 14
Completed | 1 | 1
Not Completed | 26 | 13
Not completed — Lack of Efficacy | 17 | 6
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Terminated participation | 6 | 2
Not completed — Seek alternative treatment | 2 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Then Secukinumab: Placebo via subcutaneous injection using 2 prefilled syringes at Weeks 0, 1, 2, 3, 4.
  Thereafter through Week 16, the first 36 patients assessed at baseline received placebo Q4W, while the remaining 5 patients received a higher dosing schedule of placebo Q2W.
  Starting at Week 16, all subjects received secukinumab 300 mg. Patients initially randomized to placebo Q4W or the higher dosing placebo Q2W received secukinumab 300 mg Q4W from Week 16 to Week 20, followed by every 4 weeks until Week 48 or every 2 weeks through Week 48 for the higher dosing schedule.
- Secukinumab Only: Secukinumab (300 mg) via subcutaneous injection using 2 prefilled syringes at Weeks 0, 1, 2, 3, 4.
  Thereafter through Week 16, the first 36 patients assessed at baseline received secukinumab 300 mg Q4W, while the remaining 5 patients received a higher dosing schedule of secukinumab 300 mg Q2W.
  Starting at Week 16, all subjects received secukinumab 300 mg. Patients initially randomized to secukinumab 300 mg Q4W or the higher dosing secukinumab 300 mg Q2W continued to receive their respective dosages through Week 48.
- Total: Total of all reporting groups
Arm/Group | Placebo Then Secukinumab | Secukinumab Only | Total
Number analyzed (Participants) | 14 | 27 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (15.9) | 38.3 (13.8) | 36.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 8 | 15 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 14 | 24 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 10 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 6 | 14 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Eczema Area and Severity Index (EASI) score [Mean (Standard Deviation); unit: units on a scale] — The EASI index assigns proportionate values to 4 body regions. Each region is assigned a score of 0 to 3, indicating none, mild, moderate, and severe clinical expression. The percentage of area involved is also assigned an eruption proportional score from 0 to 6. The total body score for each body region is obtained by multiplying the sum of the severity scores by the area score, then multiplying the result by the constant weighted value assigned to that body region. The sum of these scores gives the EASI total from 0-72, with higher score indicating more severity.
  units on a scale | 29.9 (12.6) | 29.0 (12.0) | 29.3 (12.04)
SCORing Atopic Dermatitis (SCORAD) score [Mean (Standard Deviation); unit: units on a scale] — SCORing Atopic Dermatitis -The intensity part of the SCORAD index consists of six items: erythema, edema⁄papulation, excoriations, lichenification, oozing⁄crusts and dryness. Each item graded on a scale 0-3. The subjective items include daily pruritus and sleeplessness, graded on a 10-cm visual analogue scale, with maximum subjective score 20. SCORAD full score is 0-103, with higher score indicating more symptoms.
  units on a scale | 63.3 (14.1) | 65.0 (12.7) | 64.4 (13.0)
IgE level [Mean (Standard Deviation); unit: kU/L] — Intrinsic Atopic Dermatitis IgE =< 500 kU/L; Extrinsic Atopic Dermatitis, IgE > 500 kU/L
  kU/L | 3424 (3509) | 5101 (11157) | 4555.8 (9348.9)

OUTCOME MEASURES:

1. Primary Outcome: Fold-Change in Epidermal Thickness of Lesional Skin
Description: Epidermal hyperplasia assessed using change in epidermal thickness at week 16 as compared to baseline
Time Frame: at Week 16
Population: Data only for those that returned for week 16 visit
Measure: Mean (Standard Error); unit: fold-change
Groups:
- Placebo Then Secukinumab for Extrinsic AD; Placebo Then Secukinumab for Intrinsic AD: Placebo via subcutaneous injection using 2 prefilled syringes at Weeks 0, 1, 2, 3, 4.
  Thereafter through Week 16, the first 36 patients assessed at baseline received placebo Q4W, while the remaining 5 patients received a higher dosing schedule of placebo Q2W.
  Starting at Week 16, all subjects received secukinumab 300 mg. Patients initially randomized to placebo Q4W or the higher dosing placebo Q2W received secukinumab 300 mg Q4W from Week 16 to Week 20, followed by every 4 weeks until Week 48 or every 2 weeks through Week 48 for the higher dosing schedule.
- Secukinumab Only for Extrinsic AD; Secukinumab Only for Intrinsic AD: Secukinumab (300 mg) via subcutaneous injection using 2 prefilled syringes at Weeks 0, 1, 2, 3, 4.
  Thereafter through Week 16, the first 36 patients assessed at baseline received secukinumab 300 mg Q4W, while the remaining 5 patients received a higher dosing schedule of secukinumab 300 mg Q2W.
  Starting at Week 16, all subjects received secukinumab 300 mg. Patients initially randomized to secukinumab 300 mg Q4W or the higher dosing secukinumab 300 mg Q2W continued to receive their respective dosages through Week 48.
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 7 | 3 | 14 | 8
fold-change | 1.15 (1.22) | 1.5 (1.3) | 1.18 (1.15) | -1 (1.15)

2. Secondary Outcome: Fold-Change in K16 Expression of Lesional Skin
Description: Epidermal hyperplasia assessed using change in the epidermal proliferation marker Ki67 at week 16 as compared to baseline. Staining quantification was performed with ImageJ 1.42
Time Frame: at Week 16
Measure: Mean (Standard Error); unit: fold-change
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 7 | 3 | 14 | 8
fold-change | 1.14 (1.89) | -3.96 (2.33) | 1.36 (1.56) | -1.3 (1.84)

3. Secondary Outcome: Number of Patients With SCORAD-50
Description: The proportion of patients who achieve an improvement of 50% or greater from their Baseline objective SCORAD up to week 52. SCORing Atopic Dermatitis (SCORAD) -The intensity part of the SCORAD index consists of six items: erythema, edema⁄papulation, excoriations, lichenification, oozing⁄crusts and dryness. Each item graded on a scale 0-3. The subjective items include daily pruritus and sleeplessness, graded on a 10-cm visual analogue scale, with maximum subjective score 20. SCORAD full score is 0-103, with higher score indicating more symptoms.
Time Frame: Week 4, Week 16, Week 32, Week 52
Population: data for participants who returned for the respective week visit
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 8 | 5 | 17 | 10
Participants
  Week 4 | 0 | 0 | 2 | 0
  Week 16: number analyzed (Participants) | 7 | 3 | 14 | 8
  Week 16 | 0 | 0 | 3 | 2
  Week 32: number analyzed (Participants) | 1 | 2 | 1 | 2
  Week 32 | 0 | 0 | 0 | 1
  Week 52: number analyzed (Participants) | 1 | 0 | 0 | 1
  Week 52 | 1 | 0 | 0 | 1

4. Secondary Outcome: Number of Patients Who Achieve EASI-50 Score
Description: The proportion of patients who achieve an improvement of 50% or greater from their Baseline EASI score up to week 52. The EASI index assigns proportionate values to 4 body regions. Each region is assigned a score of 0 to 3, indicating none, mild, moderate, and severe clinical expression. The percentage of area involved is also assigned an eruption proportional score from 0 to 6. The total body score for each body region is obtained by multiplying the sum of the severity scores by the area score, then multiplying the result by the constant weighted value assigned to that body region. The sum of these scores gives the EASI total from 0-72, with higher score indicating more severity.
Time Frame: Week 4, Week 16, Week 32, Week 52
Population: data for participants who returned for the respective week visit
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 8 | 5 | 17 | 10
Participants
  Week 4 | 0 | 0 | 1 | 0
  Week 16: number analyzed (Participants) | 7 | 3 | 14 | 8
  Week 16 | 0 | 1 | 3 | 4
  Week 32: number analyzed (Participants) | 1 | 2 | 1 | 2
  Week 32 | 0 | 2 | 0 | 1
  Week 52: number analyzed (Participants) | 1 | 0 | 0 | 1
  Week 52 | 1 | 0 | 0 | 1

5. Secondary Outcome: Number of Patients With Static Investigator's Global Assessment (IGA) Score 0 or 1
Description: The proportion of patients who achieve a score of "clear-0" or "almost clear-1" in the static IGA score at Week 16 as compared to Baseline. The static IGA score represents an overall static evaluation of dermatitis, performed by the investigator at each visit. It utilizes a scale of 6-points; total scale ranging from 0 (clear) to 5 (very severe disease).
Time Frame: Week 16, Week 32, Week 52
Population: data for participants who returned for the respective week visit
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 8 | 5 | 17 | 10
Participants
  Week 16: number analyzed (Participants) | 7 | 3 | 14 | 8
  Week 16 | 0 | 0 | 0 | 1
  Week 32: number analyzed (Participants) | 1 | 2 | 1 | 2
  Week 32 | 0 | 0 | 0 | 0
  Week 52: number analyzed (Participants) | 1 | 0 | 0 | 1
  Week 52 | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage Change From Baseline in SCORAD Score
Description: Percentage change in SCORAD scores at Week 16 as compared to baseline. SCORing Atopic Dermatitis (SCORAD) full score is 0-103, with higher score indicating more symptoms.
Time Frame: at Week 16
Population: data for participants who returned for the week 16 visit
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 7 | 3 | 14 | 8
percentage change | -3.19 (9.92) | -27.31 (7.48) | -8.54 (6.22) | -6.11 (13.85)

7. Secondary Outcome: Percentage Change From Baseline in EASI Scores
Description: Percentage change in EASI scores at Week 16 as compared to baseline. Eczema Area and Severity Index (EASI) total score from 0-72, with higher score indicating more severity.
Time Frame: at Week 16
Population: Data analysis only for those who returned for Week 16 visit
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 7 | 3 | 14 | 8
percentage change | 5.27 (12.71) | -28.74 (15.01) | -4.96 (7.54) | -16.9 (18.92)

8. Secondary Outcome: Fold-Change in Elafin/Pi3 Level From Baseline
Description: Change of IL-17 regulated keratinocyte products assessed by a change of the mRNA gene expression levels of elafin/Pi3 at week 16 as compared to baseline
Time Frame: at Week 16
Population: Data analysis only for those who returned for Week 16 visit
Measure: Mean (Standard Error); unit: fold-change
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 7 | 3 | 14 | 8
fold-change | -1.00 (2.06) | -7.90 (2.60) | 1.3 (1.66) | -2.65 (2.00)

9. Secondary Outcome: Fold-Change in CCL20 Level
Description: Change of IL-17 regulated keratinocyte products assessed by a change of the mRNA gene expression levels of CCL20 at week 16 as compared to baseline.
Time Frame: at Week 16
Population: Data analysis only for those who returned for Week 16 visit
Measure: Mean (Standard Error); unit: fold-change
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 7 | 3 | 14 | 8
fold-change | 1.35 (1.76) | -1.38 (2.10) | 1.23 (1.48) | -1.85 (1.72)

10. Secondary Outcome: Fold-Change in CXCL1 Level
Description: Change of IL-17 regulated keratinocyte products assessed by a change of the mRNA gene expression levels of CXCL1 at week 16 as compared to baseline.
Time Frame: at Week 16
Population: Data analysis only for those who returned for Week 16 visit
Measure: Mean (Standard Error); unit: fold-change
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 7 | 3 | 14 | 8
fold-change | 1.12 (1.71) | -2.72 (2.02) | 1.31 (1.45) | -1.38 (1.67)

11. Secondary Outcome: Fold-Change in S100A7 Level
Description: Change of IL-17 regulated keratinocyte products assessed by a change of the mRNA gene expression levels of S100A7 at week 16 as compared to baseline.
Time Frame: at Week 16
Population: Data analysis only for those who returned for Week 16 visit
Measure: Mean (Standard Error); unit: fold-change
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 7 | 3 | 14 | 8
fold-change | -1.13 (1.83) | -5.25 (2.24) | 1.43 (1.52) | -2.59 (1.79)

12. Secondary Outcome: Fold-Change in A8 Level
Description: Change of IL-17 regulated keratinocyte products assessed by a change of the mRNA gene expression levels of A8 at week 16 as compared to baseline
Time Frame: at Week 16
Population: Data analysis only for those who returned for Week 16 visit
Measure: Mean (Standard Error); unit: fold-change
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 7 | 3 | 14 | 8
fold-change | -1.32 (2.12) | -9.51 (2.72) | 1.51 (1.69) | -2.61 (2.1)

13. Secondary Outcome: Fold-Change in A9 Level
Description: Change of IL-17 regulated keratinocyte products assessed by a change of the mRNA gene expression levels of A9 at Week 16 as compared to baseline.
Time Frame: at Week 16
Population: data only for those who returned for week 16 visit
Measure: Mean (Standard Error); unit: fold-change
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 7 | 3 | 14 | 8
fold-change | -1.47 (0.86) | -20.03 (1.36) | 1.58 (0.6) | -2.16 (0.85)

14. Secondary Outcome: Fold-Change in A12 Level
Description: Change of IL-17 regulated keratinocyte products assessed by a change of the mRNA gene expression levels of A12 as compared to baseline
Time Frame: at Week 16
Measure: Mean (Standard Error); unit: fold-change
Arm/Group | Placebo Then Secukinumab for Extrinsic AD | Placebo Then Secukinumab for Intrinsic AD | Secukinumab Only for Extrinsic AD | Secukinumab Only for Intrinsic AD
Number analyzed (Participants) | 7 | 3 | 14 | 8
fold-change | 1.24 (2.24) | -15.06 (2.91) | 1.95 (1.76) | -2.87 (2.17)

ADVERSE EVENTS:
Time Frame: up to 52 weeks
Arm/Group | Placebo Then Secukinumab | Secukinumab Only
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/27
Other Adverse Events (participants affected / at risk) | 0/14 | 3/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Then Secukinumab (N=14) | Secukinumab Only (N=27)
Orbital Cellulitis (Infections and infestations) | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 0 | 1
Streptococcal Pharyngitis (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT02594098/Prot_SAP_000.pdf